CLINICAL TRIAL: NCT00357058
Title: Substrates Mediating Deafferentiation-Induced Enhancement of Tactile Spatial Acuity
Brief Title: Role of Brain Region Changes in Tactile (Touch) Ability Following Nerve Block
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020079; 02-N-0079
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-28

CONDITIONS: Tactile Spatial Acuity; Healthy
Keywords: Deafferentiation-Induced Plasticity; fMRI; Cortical Reorganization; Tactile Performance; Transcranial Magnetic Stimulation; Tactile Discrimination; Plasticity; Healthy Volunteer; HV; Normal Control

SUMMARY:
This study will examine the role of different brain regions in tactile (touch) ability after application of a tourniquet (inflated blood pressure cuff). When the forearm is deprived of blood for a short period of time, tactile ability in the other hand improves. This study will try to learn what causes this improvement.

Healthy normal volunteers are eligible for this study. Candidates will have a brief medical history and physical examination.

Volunteers will undergo two experiments, described below, that involve the following procedures:

* Ischemic nerve block - A blood pressure cuff is inflated for 35-40 minutes around the elbow area (also around the calf for Experiment 2 - see below). The resulting numbness, tingling, loss of muscle strength, and discoloration of the forearm and hand disappear within minutes after the cuff is deflated.
* Magnetic resonance imaging (MRI) - This test uses a magnetic field and radio waves instead of X-rays to produce images of brain structure and function. The volunteer lies on a stretcher that is moved into the scanner (a cylinder containing a strong magnet), wearing earplugs to protect the ears from loud thumping noises that occur with electrical switching of radio frequency circuits. The subject can communicate with an investigator by intercom at all times during the scan.
* Transcranial magnetic stimulation (TMS) - An insulated wire coil is placed on the patient's scalp. A brief electrical current passes through the coil, creating a magnetic pulse that travels through the scalp and skull and causes small electrical currents in the outer part of the brain. The stimulation may cause muscle hand or arm twitching or transient tingling in the forearm, head or face muscles.
* Tactile spatial acuity testing - The subject's left arm is placed in a cast and the left index finger is immobilized for this test which involves identifying the direction of grooves applied to the finger.

Experiment 1

This experiment measures changes in tactile acuity and brain activation following cuff inflation. The subject lies in the MRI scanner, with the left arm immobilized. Tactile acuity is measured repetitively at the left index finger during placement and inflation of a pressure cuff around the right forearm. The experiment consists of two sessions with the cuff around the forearm and one with the cuff around the calf and lasts from 90 minutes to 2 hours.

Experiment 2

This experiment measures changes in tactile acuity linked to TMS stimulation. The subject sits in an armchair with the left arm immobilized. Tactile acuity is measured repetitively at the left index finger during placement and inflation of a pressure cuff around the right forearm. In addition, TMS pulses (about one pulse per second) are delivered at different locations over the right side of the head for up to 30 minutes. The experiment consists of 10 separate sessions on different days, each lasting about 1 hour.

DETAILED DESCRIPTION:
Acute deafferentation in one hand leads to improvements in tactile discriminative skills in the other, non-deafferented hand. This phenomenon, recently identified in our laboratory, represents an adaptive, behaviorally important consequence of deafferentation. It demonstrates that acute loss of sensory input from one hand results in rapid improvement of skills in the remaining hand. The first experiment in this protocol seeks to identify cortical regions activated in association with this improvement in tactile spatial acuity. In the second experiment, we will determine the effects of transient inactivation of focal cortical regions on this behavioral gain. While the first experiment will characterize brain regions activated in association with this performance improvement, the second experiment will provide information on the functional role of these regions. Understanding the substrates that mediate this behavioral gain may be important for the design of strategies to enhance them.

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal volunteers who are willing and able to remain relaxed and immobile during active scans, for a period of up to 2 hours.

EXCLUSION CRITERIA:

Subjects with: metal in the cranium except for crowns or fillings in mouth and permanent metal dental braces, metal fragments from occupational exposure or surgical clips in or near the brain.

Subjects with eye, blood vessel, cochlear or eye implants, with increased intracranial pressure as evaluated by clinical means, with cardiac or neural pacemakers, intracardiac lines and/or implanted medication pumps.

Subjects with large hemorrhagic or brain stem stroke.

Subjects with multiple cerebral lesions with residual deficits.

Subjects with history of head injury with loss of consciousness.

Subjects with history of severe alcohol or drug abuse or psychiatric illness.

Subjects with unstable cardiac dysrhythmia or unresponsive arterial hypertension (greater than 160/100 mmHg).

Subjects with history of hyperthyroidism or individuals receiving drugs acting primarily on the central nervous system or disorders of the blood coagulation system.

Subjects with excessive callus at their fingers.

Preganant women will be excluded from the study.

SUBJECTS DISCONTINUATION CRITERIA:

Subject's poor compliance with protocol evaluations or examinations and subject's request to withdraw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2001-12-12; Study Completion 2007-12-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Allard T, Clark SA, Jenkins WM, Merzenich MM. Reorganization of somatosensory area 3b representations in adult owl monkeys after digital syndactyly. J Neurophysiol. 1991 Sep;66(3):1048-58. doi: 10.1152/jn.1991.66.3.1048. PMID 1753275